CLINICAL TRIAL: NCT05845099
Title: Assessment of Microbial Adherence and Patients' Satisfaction in Conventional and Digital 3D Printed Complete Removable Dentures: A Cross Over Randomized Controlled Clinical Trial
Brief Title: Conventional Versus Digital 3D Printed Complete Removable Dentures
Acronym: CRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M Refai, Lecturer of Oral and Maxillofacial Prosthodontics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-Re IR112224
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Denture, Complete
Keywords: 3D printing; CAD/CAM; Complete dentures

STUDY DESIGN:
Intervention Model Description: double blind single center crossover design
Who Masked: Participant, Care Provider, Investigator
Masking Description: neither the patients nor the operator know which type of denture will be inserted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polymethyl Methacrylate-Based Complete Removable Dentures. (Active Comparator): The patient will be provided by a CRD to restore his missing teeth which will be manufactured by heat curing processing technique
  Interventions: Device: Polymethyl Methacrylate-Based Complete Removable Dentures.
- Photopolymerized Methacrylate- Based Complete Removable Dentures. (Experimental): The patient will be provided by a CRD to restore his missing teeth which will be manufactured by 3D-printed (Digital Light Processing).
  Interventions: Device: Photopolymerized Methacrylate- Based Complete Removable Dentures.

INTERVENTIONS:
Device: Polymethyl Methacrylate-Based Complete Removable Dentures. — The patients will receive Complete Removable Dentures processed by Heat cured acrylic resin.
  Other Names: Complete Removable Denture manufacturing
  Arms: Polymethyl Methacrylate-Based Complete Removable Dentures.
Device: Photopolymerized Methacrylate- Based Complete Removable Dentures. — The patients will receive a 3D-printed removable denture digitally manufactured using a 3d printer device with light polymerized resin.
  Other Names: 3D printed Removable Denture manufacturing
  Arms: Photopolymerized Methacrylate- Based Complete Removable Dentures.

SUMMARY:
The study is a crossover, randomised, controlled clinical trial that will compare and evaluate patients' satisfaction and oral microbiota proliferation in two groups. Group I: Conventionally manufactured CRD Group II: 3D-printed (three-dimensionally printed) CAD/CAM (computer-aided design/computer-aided manufacturing) manufactured CRD, The participants will be selected according to inclusion and exclusion criteria and will be randomly allocated into both groups and then shuffled to the other group using the Research Randomizer Program.

DETAILED DESCRIPTION:
The study will be performed at the outpatient clinic of the Oral and Maxillofacial Prosthodontics Department, Faculty of Dentistry, Ain Shams University. Eleven edentulous male patients will be selected and recruited for this clinical trial after the informed consent provided by Faculty of Dentistry Ain Shams University-Research Ethics Committee (FDASU-REC) is assigned. They will be rehabilitated with Conventional and 3D-printed CAD-CAM (computer-aided design/computer-aided manufacturing) CRD. Participants will be randomly assigned to receive either Conventional or 3D-Printed CAD/CAM-manufactured CRD for three months before crossing over to the other set. care provider , investigator and participants will be blinded to the group allocation. Outcomes will be evaluated, including patient satisfaction with dentures and oral microbial adherence. The outcomes will be measured at baseline and at 1 and 3 months. The obtained data will be recorded, tabulated, and statistically analyzed using the appropriate tests for comparison between each group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been completely edentulous in both jaws (maxilla and mandible) for at least a year and require treatment with complete dentures.
2. The age of patients ranges from 45 to 60 years old.
3. Patients with a Class I maxillo-mandibular relationship.
4. Patients with adequate inter-arch space.
5. Patients with good neuromuscular control.
6. Patients without any temporomandibular joint disorder.

Exclusion Criteria:

1. Patients with any oral diseases that may affect complete denture construction.
2. Patients with bad oral hygiene.
3. Patients with oral parafunctional habits.
4. Hysterical patients.
5. Patients will undergo or have previously received chemotherapy or radiotherapy.
6. Smokers or drug- addicted patients

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will include male patients only as old female patients can suffer from menopause and decreased immunity
Enrollment: 20 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Assessment of oral microorganism proliferation by talking swab from | 3 months
  Assessment of oral microorganism proliferation by talking swab from the internal surface of both types of CRD to asses the affinity of oral microorganisms.

SECONDARY OUTCOMES:
Evaluation of patients' satisfaction with both types of the Complete Removable Dentures | 3 months
  Evaluation of patients' satisfaction with both types of the Complete Removable Dentures by using Patient's Denture Assessment questionnaire (PDA) and interpreting it by using Likert scale (higher score (scale no.5) indicates good outcome and lower score (scale no.1)indicates bad outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Omnia MS Refai, PHD, Study Chair — lecturer of Oral and Maxillofacial Prosthodontics, Faculty of Dentistry , Ain Shams University; Heba RF Elsarrif, PHD, Study Director — Lecturer of Oral and Maxillofacial Prosthodontics College of oral and dental surgery Misr University for science and technology
Locations (1):
- Faculty of Dentistry, Ain shams University, Cairo, Egypt

REFERENCES:
- [Background] Srinivasan M, Kalberer N, Fankhauser N, Naharro M, Maniewicz S, Muller F. CAD-CAM complete removable dental prostheses: A double-blind, randomized, crossover clinical trial evaluating milled and 3D-printed dentures. J Dent. 2021 Dec;115:103842. doi: 10.1016/j.jdent.2021.103842. Epub 2021 Oct 9. PMID 34637889
- [Background] Baba NZ, AlRumaih HS, Goodacre BJ, Goodacre CJ. Current techniques in CAD/CAM denture fabrication. Gen Dent. 2016 Nov-Dec;64(6):23-28. PMID 27814252